CLINICAL TRIAL: NCT03352310
Title: Umbilical Cord Blood Mononuclear Cell Bank in Hong Kong and Treatment of Neonatal Cerebral Ischemia and Anemia - Part IV Clinical Trial
Brief Title: Feasibility and Safety of Umbilical Cord Blood Transfusion in the Treatment of Neonatal Cerebral Ischemia and Anemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mononuclear Therapeutics Ltd. (Industry)
Collaborators: Chinese University of Hong Kong (Other); China Spinal Cord Injury Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB-HIEA-01
Record Dates: First submitted 2017-11-15; First posted 2017-11-24 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Hypoxia Neonatal; Cerebral Ischemia of Newborn; Anemia, Neonatal
Keywords: umbilical cord blood
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum; Anemia, Neonatal | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Study Group - autologous umbilcial cord blood transfusion
  Control Group - standard care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): autologous UCB transfusion
  Interventions: Biological: autologous umbilical cord blood (UCB)
- Control Group (Other): standard care
  Interventions: Procedure: standard care

INTERVENTIONS:
Biological: autologous umbilical cord blood (UCB) — autologous UCB transfusion to the newborn infants presence of HIE and/or anemia within 48 hours after the birth
  Arms: Study Group
Procedure: standard care — standard care procedure to the newborn infants presence of HIE and/or anemia
  Arms: Control Group

SUMMARY:
The study is to investigate the feasibility and safety of autologous umbilical cord blood transfusion to treat the newborn infants with presence of clinical indications of neonatal hypoxic-ischemia encephalopathy (HIE) and anemia. Umbilical cord blood (UCB) is collected following labor and is transfused intravenously within 48 hours after the birth. Newborn infant without UCB available recieves the standard care will be enrolled as control group.

Following the autologous UCB transfusion in the study group or standard care in the control group, HIE subjects will be followed for 2 years for survival and neurodevelopmental outcomes and anemia subjects will be followed for 6 months to assess the survival and change of hematocrit and hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* evidence of asphyxiation, defined by 5-minute Apgar score ≤ 5;
* evidence of HIE, defined by UCB pH <7.15 or base excess ≤ 10mM;
* subjects with HIE confirmed by clinical features and initial investigations;
* subjects with evidence of anemia, defined by hematocrit < 40% or hemoglobin ≤ 13g/dL within the first 96 hours of life;
* obtain the informed consent from parents

Exclusion Criteria:

* congestive cardiac failure;
* microcephaly, anencephaly, encephalocele, or other abnormality
* conjoint twins;
* chromosomal disorders
* fetal alcohol syndrome
* spinal bifida or other neural tube defects
* subjects have other neurological deficit conditions
* polycythemia
* congenital hematological malignancy
* investigator decision

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
HIE: Mortality | 6 months
  Mortality Rate of the HIE Subjects
Anemia: Change from Baseline Hematocrit | 48 hours, 1 week, 3 months, 6 months
  Change from Baseline Hematocrit of the Anemia Subjects

SECONDARY OUTCOMES:
HIE: HINE | 6 months, 1 year and 2 years
  Hammersmith Infant Neurological Examination (HINE) of the HIE Subjects
HIE: HNNE | -1 day, 3 months (before discharge)
  Hammersmith Neonatal Neurological Examination (HNNE) of the HIE Subjects
HIE: GMDS | 6 months, 1 year and 2 years
  Griffiths Mental Development Scale (GMDS) of the HIE Subjects
HIE: CBCL | 2 years
  Child Behavior Checklist for Attention Deficit of the HIE Subjects
HIE: Q-CHAT | 2 years
  Quantitative Checklist for Autism in Toddlers of the HIE Subjects
Anemia: hemoglobin | 48 hours, 1 week, 3 months and 6 months
  Change from Baseline hemoglobin of the Anemia Subjects
Anemia: Oxygenation level | 48 hours, 1 week
  Change from Baseline SpO2 of the Anemia Subjects
Anemia: Oxidative Stress Level | 48 hours, 1 week, 3 months, and 6 months
  Change of Baseline Isoprostane of the Anemia Subjects
Anemia: Requirements of Packed Cell Transfusion | 6 months
  Frequency of Requirements of Packed Cell Transfusion by the Anemia Subjects

OTHER OUTCOMES:
Incidence of Adverse Event | 2 years
  Safety outcomes are Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided